CLINICAL TRIAL: NCT02846454
Title: Investigating the Effects of a Composite Drink of Inulin and Arabinoxylan on Satiety, Energy/Food Intake and Changes in the Human Gut Microbiota
Brief Title: Effects of Inulin and Arabinoxylan on Satiety, Energy/Food Intake and Changes in the Human Gut Microbiota
Acronym: MIXSAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Dr Daniel Commane, Principal Investigator, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UReading
Record Dates: First submitted 2016-06-20; First posted 2016-07-27 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Inulin; arabinoxylan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- inulin (Experimental): Investigating the satiating effects of consuming 4g/d inulin (Fruitafit IQ by CHIMAB)
  Interventions: Other: inulin
- non inulin and arabinoxylan (No Intervention): investigating the satiating effects of a control drink (2.6g/d maltodextrin)
- arabinoxylan (Experimental): Investigating the satiating effects of consuming 4g/d arabinoxylan (Medium Chain Naxus, BioActor b.v)
  Interventions: Other: arabinoxylan

INTERVENTIONS:
Other: inulin — Investigate the satiating effects of consuming 4g/d inulin in 2 daily doses of 2g
  Other Names: Inulin (Fruitafit IQ)
  Arms: inulin
Other: arabinoxylan — Investigate the satiating effects of consuming 4g/d arabinoxylan in 2 daily doses of 2g
  Other Names: arabinoxylan (Naxus)
  Arms: arabinoxylan

SUMMARY:
This proposed randomized, double blinded 12 week crossover human feeding study aims to investigate the effects of consuming a composite drink of inulin and arabinoxylan on satiety by measuring appetite biomarkers such as subjective satiety, energy/food intake and changes in the human gut microbiota in healthy weight males (22 to 24.9kg/m2)

DETAILED DESCRIPTION:
Research that focuses on the mechanisms involved in appetite regulation is topical given the emergence of the worldwide obesity epidemic. Understanding the physiological processes associated with the onset of obesity is essential for the development of effective anti-obesity strategies. There is evidence that people who consume a diet high in non-starch polysaccharides (NSPs) have a lower body mass index (BMI) than those that do not.

A 2009 review of fibre and satiety by Bridget Benelam, 2009 focused on different types of fibre and the significant impact they may have on satiety and/or energy intake, through fermentation of fibre such as non starch polysaccharides in the colon by gut bacterial groups such as Bifidobacterium. non starch polysaccharides and other fibre sources are poorly digested by human enzymes in the small intestine but are degraded by large groups of bacteria in the large bowel. One of the beneficial outcomes of this fermentation of fibre that gut bacteria produce of metabolites called short chain fatty acids (SCFA) thought to affect appetite regulation by stimulating production of satiety hormones that can help you feel full. Acetate and propionate are two of these metabolites highlighted as potential mediator of satiety.

Some fibres are called prebiotics as they act as selective sources for beneficial gut bacteria. However Western populations do not consume natural prebiotics in high quantities in their diet and the overall intake of fibre is also low. Therefore, in this study, the investigators aim to utilise a mixture of prebiotics in order to increase the growth and/or activity of commensal gut bacteria and SCFA production in human volunteers and to assess the effects of consumption on satiety.

Testing the impact of a composite mix of inulin and arabinoxylan in a human study will help determine the effect it has on appetite regulation, ad libitum food intake, SCFA production, anthropometric measurements, cognitive state (e.g. mood) and composition of the gut microbiota.

The study design is a 12 week randomized, human feeding study, with a crossover design testing a composite mix of inulin and arabinoxylan against an equivalent energy matched (kcal) maltodextrin control drink in 33 healthy weight (22 to 24.9kg/m2) males aged between 21-55. Volunteers will be enrolled to treatment or placebo for four weeks, with a four week wash out before the crossover. the primary endpoint, satiety following a test meal challenge will be measured on four occasions throughout the study. Anthropometry measures, dietary intake, body weight and blood pressure will be monitored throughout the study. Faecal and urine will be collected at baseline and at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 21-55 years old
* Body Mass Index (BMI) 19.5-24.5kg/m2
* Overall healthy
* Weight Stable (<3 kg change in the past 4 months, before the trial).

Exclusion Criteria:

* Smokers
* drink more than 28 units of alcohol per week (i.e. not more than 14 pints of beer or 28 small glasses of wine)
* Restricted diet such as weight loss, vegetarian/vegan or taking dietary supplements such as prebiotics (such as oligosaccharides ie Fructo-oligosaccharides (FOS), galacto-oligosaccharides (GOS) or probiotics (ie Actimel)), not eating breakfast and >25g/d dietary fibre consumption as well as those with food allergies
* Gastrointestinal procedure or surgery in the past three months.
* Gastrointestinal disorders: celiac disease, Intestinal Bowel Disease (IBD), irritable bowel syndrome (IBS), chronic constipation, diverticulitis or a history of chronic constipation, diarrhoea, or other chronic gastrointestinal complaints
* Disorders of swallowing, severe dysphagia to food or pills.
* Appetite modulator drugs: orlistat, sibutramine, rimonabant.
* Mood disorder medications: antidepressants, lithium.
* Chronic metabolic conditions: diabetes, hepatic disease, gout, kidney, thyroid or coagulation disease.
* Psychiatric disorder: severe depression, bulimia, anorexia, schizophrenia, bipolar disorder.
* Pregnancy
* Others: oral antidiabetics, insulin, digoxin, thyroid hormones, antibiotics, steroids or immunosuppressants, recreational substances.
* Use of implanted or portable electro-mechanical device such as cardiac peacemaker or infusion pump.
* Blood donor in the past 3 months.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Effects of consuming a composite drink of inulin and arabinoxylan on subjective satiety scores | 6hrs
  The volunteers will randomized to receive either control or treatment drink and asked to consume this twice daily for 28 days, followed by a 28 day washout, the alternate drink will then be consumed for a further 28 days. Visual analogue scale will be used to measure subjective satiety scores during 4 half day study days lasting 6hrs at the beginning and end of each treatment period at a designated nutrition unit (Hugh Sinclair Nutrition unit, Reading University).

SECONDARY OUTCOMES:
Effects of consuming a composite drink of inulin and arabinoxylan on energy intake | 6hr
  Energy intake will be measured during each of the 4 study days. A test meal of cheese and tomato pizza will be given ad libitum as a lunch meal and the energy intake (KJ) will be measured by weighing the food before and after consumption.
Effects of consuming a composite drink of inulin and arabinoxylan on anthropometric measurements | 12 weeks
  In order to see if consumption of inulin and arabinoxylan have impacted anthropometric measurements, these will also be taken at the beginning of each of the 4 study days including height (m), weight (kg), waist and hip circumference (cm).
Effects of consuming a composite drink of inulin and arabinoxylan on mediating changes in gut microbiota | 28 days
  To assess the changes in faecal bacteria populations using fluorescent in situ hybridisation (FISH) will be used in which molecular probes target 16S ribosomal ribonucleic acid (rRNA),labelled with the fluorescent Cy3 dye (Sigma Aldrich Ltd., Poole, Dorset, UK) and as previously described by Martín-Peláez S et al 2008
Effects of consuming a composite drink of inulin and arabinoxylan on the production of short chain fatty acid production. | 28 days
  Analysis of SCFA production will be measured in millimolar (mM) by High Performance Liquid Chromotography (HPLC) and analysis using quantitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Proven, PhD, Study Chair — Ethics committee Co-ordinator
Locations (1):
- Mr Daniel commane, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin-Pelaez S, Gibson GR, Martin-Orue SM, Klinder A, Rastall RA, La Ragione RM, Woodward MJ, Costabile A. In vitro fermentation of carbohydrates by porcine faecal inocula and their influence on Salmonella Typhimurium growth in batch culture systems. FEMS Microbiol Ecol. 2008 Dec;66(3):608-19. doi: 10.1111/j.1574-6941.2008.00610.x. PMID 19049655
- [Background] Benelam, B. Satiation, satiety and their effects on eating behaviour., 2009. British Nutrition Foundation, 34(2).
- [Derived] Collins SM, Gibson GR, Stainton GN, Bertocco A, Kennedy OB, Walton GE, Commane DM. Chronic consumption of a blend of inulin and arabinoxylan reduces energy intake in an ad libitum meal but does not influence perceptions of appetite and satiety: a randomised control-controlled crossover trial. Eur J Nutr. 2023 Aug;62(5):2205-2215. doi: 10.1007/s00394-023-03136-6. Epub 2023 Apr 12. PMID 37046122